CLINICAL TRIAL: NCT06551428
Title: The Sleep Stress Connection: Investigating How Sleep Quality Affects Mental and Physical Health
Brief Title: The Effect of Sleep Quality on Mental and Physical Health
Status: Not yet recruiting | Type: Observational
Sponsor: Ahmed Ali Mohammed Torad (Other)
Responsible Party: Sponsor-Investigator, Ahmed Ali Mohammed Torad, Lecturer at department of the basic sciences, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Other Study IDs: KFSIRB200-267
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Issue; Physical Stress
Keywords: Sleep and mental health; Stress-sleep connection; Mental health and sleep; Sleep disorders and health impact; Sleep and stress effects; Sleep impact on Physical health; Sleep quality
MeSH Terms: conditions — Psychological Well-Being; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- university students between age of 15 and 35

SUMMARY:
This study aimed to explore the relationship between sleep quality and its impact on mental and physical health, particularly in the context of stress.

A mixed methods approach will be used including:

a pre-test questionnaire and physiological measurements that depend on scales for measuring to assess sleep patterns: DASS21, fatigue assessment scale, Epworth sleeping scale, and SF-12 health survey scoring.

All of that will highlight the importance of addressing sleep quality as a crucial factor in promoting overall well-being.

DETAILED DESCRIPTION:
This study aims to explore the relationship between sleep quality and its impact on mental and physical health, particularly in the context of stress.

A mixed methods approach will be used including: a pre-test questionnaire and physiological measurements that depend on scales for measuring to assess sleep patterns: DASS21, fatigue assessment scale, Epworth sleeping scale, and SF-12 health survey scoring.

All of that will highlight the importance of addressing sleep quality as a key factor in promoting overall well-being.

In conclusion, understanding the intricate relationship between sleep quality, stress, and mental and physical health is vital for promoting holistic well-being, developing effective interventions, and improving health outcomes at individual, community, and societal levels. By recognizing the significance of this research, we can work towards creating a healthier and more resilient population.

ELIGIBILITY:
Inclusion Criteria:

-university students between the ages of 18 and 35.

Exclusion Criteria:

* People with diseases and conditions can significantly affect sleep quality, cause fatigue, and impact mental and physical health along with relevant medications that might exacerbate these issues:

Diseases and conditions:

* Restless Legs Syndrome (RLS)
* Bipolar Disorder
* Fibromyalgia:
* Parkinson's Disease
* Multiple Sclerosis (MS)
* Thyroid Disorders

Medication:

* Sleep aids
* antidepressants
* diuretics
* antihistamines
* hormonal medications
* blood pressure medications

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: kafrelsheikh university students
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Stress | Week
  Measurement tool: THE DASS-21 scale
  Unit of measurement:The DASS-21 (Depression, Anxiety, and Stress Scale - 21 items) measures psychological distress across three domains: depression, anxiety, and stress. Each of the three scales consists of 7 items, and respondents rate their experience over the past week on a 4-point Likert scale
  The scores for each domain are summed to provide a total score, which can then be categorized into different severity levels (normal, mild, moderate, severe, and extremely severe) based on specific cutoff points. Each of the three domains is measured separately, and the resulting scores are typically reported as a total score for each domain.
Sleep quality | Week
  Measurement tool:epwoth sleepiness sclae (ESS).
  Unit of measurement:
  The **Epworth Sleepiness Scale (ESS)** is used to assess daytime sleepiness. It consists of 8 scenarios, and respondents rate their likelihood of dozing off in each situation on a scale from 0 to 3:
  The total score is obtained by summing the scores for all 8 items, resulting in a score that can range from **0 to 24**. Higher scores indicate greater levels of daytime sleepiness. The following cutoff values are often used to interpret the results:
  These scores help in identifying individuals who may require further evaluation for sleep disorders.
Mental and physical health | 4 weeks
  Measurement tool:SF-12 health survey scoring.
  Unit of measurement:
  The SF-12 health survey scoring uses a unitless scale to measure health-related quality of life. The scores range from 0 to 100, with higher scores indicating better health status. The survey assesses physical and mental health across various dimensions but does not assign specific units of measurement like inches or pounds; instead, it provides a standardized score reflecting overall health.
Fatigue | Week
  Measurement tool: fatigue assessment scale.
  Unit of measurement:
  Based on subjective rating"numerical scale"

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali Torad, PhD, lecturer, Principal Investigator — Faculty of physical therapy Kafrelsheikh university; Tamer Mohamed El-Saeed, PhD, associate professor, Study Director — Cairo University; Reda Fathi Elbosaty, Bachelor student, Principal Investigator — Faculty of physical therapy, kafrelsheikh university; Noran Abdallah Essa, Bachelor student, Principal Investigator — Faculty of physical therapy, kafrelsheikh university
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request from the principal investigator.

REFERENCES:
- [Background] Scott AJ, Webb TL, Martyn-St James M, Rowse G, Weich S. Improving sleep quality leads to better mental health: A meta-analysis of randomised controlled trials. Sleep Med Rev. 2021 Dec;60:101556. doi: 10.1016/j.smrv.2021.101556. Epub 2021 Sep 23. PMID 34607184
- [Background] Irish LA, Kline CE, Gunn HE, Buysse DJ, Hall MH. The role of sleep hygiene in promoting public health: A review of empirical evidence. Sleep Med Rev. 2015 Aug;22:23-36. doi: 10.1016/j.smrv.2014.10.001. Epub 2014 Oct 16. PMID 25454674
- [Background] Uccella S, Cordani R, Salfi F, Gorgoni M, Scarpelli S, Gemignani A, Geoffroy PA, De Gennaro L, Palagini L, Ferrara M, Nobili L. Sleep Deprivation and Insomnia in Adolescence: Implications for Mental Health. Brain Sci. 2023 Mar 28;13(4):569. doi: 10.3390/brainsci13040569. PMID 37190534
- [Background] Sovold LE, Naslund JA, Kousoulis AA, Saxena S, Qoronfleh MW, Grobler C, Munter L. Prioritizing the Mental Health and Well-Being of Healthcare Workers: An Urgent Global Public Health Priority. Front Public Health. 2021 May 7;9:679397. doi: 10.3389/fpubh.2021.679397. eCollection 2021. PMID 34026720